CLINICAL TRIAL: NCT00444132
Title: Clopidogrel Reloading in Clopidogrel Resistant Patients With ACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3621-SM-CTIL
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Clopidogrel Non-Responsiveness
Keywords: clopidogrel; platelets; acute coronary syndrome; percutaneous coronary intervention
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

INTERVENTIONS:
Drug: clopidogrel

SUMMARY:
Laboratory clopidogrel resistance is associated with adverse atherothrombotic events in patients with coronary artery disease. In the proposed study we wish to prospectively assess the effect of reloading with 600 mg clopidogrel, and administer maintenance treatment with clopidogrel 150 mg/day for one month in a group of acute myocardial infarction (AMI) patients who demonstrate non-responsiveness to clopidogrel.

DETAILED DESCRIPTION:
Prior studies have demonstrated significant variability in platelet response to clopidogrel in patients with coronary artery disease (CAD). Up to 25% of patients have been shown to be non-responders to a conventional dose of clopidogrel. This phenomenon has been associated with higher incidence of recurrent cardiovascular (CVS) adverse events in patients with acute coronary syndrome (ACS), and higher incidence of peri-procedural myocardial damage, thrombotic complications, and ischemic events in patients undergoing elective percutaneous coronary intervention (PCI). Both the ex-vivo anti-platelet effect and the clinical benefit of clopidogrel are dose related. Moreover, in patients sustaining ACS while on maintenance clopidogrel treatment, reloading with 600 mg clopidogrel, resulted in further reduction in platelet aggregation, although the patients were not non-responders. Despite this, the effect of dose escalation has never been examined in patients resistant to clopidogrel. In the present study we wish to assess prospectively the effect of reloading with 600 mg clopidogrel, and double dose maintenance treatment (150 mg/day) for one month in acute myocardial infarction (AMI) patients who demonstrate non-respondese to clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* age equal or over 18 years
* acute coronary syndrome
* Clopidogrel non-responsive
* signed an informed consent

Exclusion Criteria:

* Bleeding disorder
* hypersensitivity to aspirin or clopidogrel
* any contraindication to anti-thrombotic or anticoagulant therapy
* active neoplastic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity

SECONDARY OUTCOMES:
recurrent ACS
stroke
death

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Matetzky, MD, Principal Investigator — Senior Physician, ICCU, Sheba Medical Center.
Locations (1):
- ICCU, Sheba Medical Center, Tel-hashomer, Ramat Gan, Israel